CLINICAL TRIAL: NCT04463355
Title: Video Discharge Instructions for Pediatric Gastroenteritis in an Emergency Department: a Randomized, Controlled Trial
Brief Title: Video Discharge Instructions for Pediatric Gastroenteritis in an Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Gonzalo Solis Garcia, Dr. Gonzalo Solís García, Principal Investigator, Hospital General Universitario Gregorio Marañon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GEA01
Record Dates: First submitted 2020-06-23; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Acute Gastroenteritis
Keywords: discharge instructions; video; acute gastroenteritis; pediatric emergency department

STUDY DESIGN:
Intervention Model Description: Open-label, parallel trial with a control group and an intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: usual verbal instructions (No Intervention): In this group, caregivers receive, after completing the test and prior to discharge, the usual verbal information and recommendations about AGE following the guidelines of the Spanish Society of Pediatric Emergencies. The instructions are always given by one of the main investigators to provide homogeneity in the information
- Intervention group: video discharge instructions (Experimental): Additionally to the verbal information, patients are shown a short 2-minute video providing the same information about AGE that would be given by verbal information.
  Interventions: Behavioral: Video discharge instructions

INTERVENTIONS:
Behavioral: Video discharge instructions — Short video (2 minutes) including information about clinical features, management and follow up of pediatric patients with acute gastroenteritis
  Arms: Intervention group: video discharge instructions

SUMMARY:
Video discharge instructions (VDI) have been suggested as a useful strategy to improve discharge instructions in pediatric emergency units. The goal of this study is to evaluate if the addition of VDI to usual verbal information improved the comprehension of information provided to caregivers of patients who consult for acute gastroenteritis (AGE). An open-label, parallel, randomized trial was designed, enrolling patients who consult for AGE. First, caregivers answer a written test concerning AGE characteristics and management. They are randomly allocated to a control group, which receives verbal discharge instructions, or to an intervention group, which additionally receives video discharge instructions. After discharge, caregivers are contacted by telephone and answer the same test. Main outcome measure is difference between test scores in the first and the second tests, secondary endpoints are how many caregivers score 5/5 on the second test, as well as rate of return visits and caregivers satisfaction with the information received.

DETAILED DESCRIPTION:
Video discharge instructions (VDI) have been suggested as a useful strategy to improve discharge instructions in pediatric emergency units. This study is designed to evaluate if the addition of VDI to usual verbal information improves the comprehension of the information provided to caregivers of patients who consult in pediatric emergency department for acute gastroenteritis (AGE). Secondary objectives are evaluating if video instructions improve satisfaction with the information received and decrease return visits.

The study is an open-label, parallel, randomized trial which takes place between June 2019 and June 2020 in the pediatric emergency department of a third-level Spanish hospital which receives 58000 emergencies annually. Up to 3 eligible patients are enrolled every shift when one of the main investigators is present. Simple, 1:1 randomization is performed using R software. Patients are randomly assigned to a group by opening sequentially numbered paper envelopes which contain the group in which the patient will be allocated, ensuring thus allocation concealment. Written informed consent is provided before trial enrollment.

Interventions

The trial is developed in three steps: an initial written test, an information phase and a second follow-up test after discharge. After enrollment, all patients fill-in a written test before discharge, which consists of 5 questions about AGE, 1 point per correct answer. Enrolled subjects are randomly assigned to the control or intervention group. In the first group of subjects (control group) caregivers receive, after completing the test and prior to discharge, the usual verbal information and recommendations about AGE following the guidelines of the Spanish Society of Pediatric Emergencies. In the second group (intervention group) patients are shown a short 2-minute video providing the same information about AGE, in addition to verbal instructions. In both groups, instructions are given by one of the main investigators in order to provide homogeneous and consistent information. Both sets of instructions explicitly include the information that had been previously asked in the test. All patients additionally receive a discharge report which includes instructions concerning aftercare treatment.

After discharge, all caregivers are contacted by telephone and asked the same 5 questions from the initial test. The questionnaire has to be completed by the same caregiver as in the previous test. This test also includes questions about subsequent visits to either emergency units or outpatient pediatric clinics and satisfaction with the information. The first telephonic contact is established 72 hours after discharge, and if unable to contact, repeated every 1-2 days up to a total of 5 days before excluding them and considering them as lost in follow-up.

Statistical Analysis The sample size was calculated to provide a statistical power of 80% at an alpha level of 5% to detect a two-tailed difference of 0.5 points between the two groups. It was calculated that with an estimated loss rate of 15% of patients between randomization and follow-up test, assuming a 1-point variance in test results based on previous studies, this statistical power would be reached by enrolling 75 patients in each group.

All randomized patients who complete both tests are included in the primary-end point analysis as part of the group in which they were randomized, following intention-to-treat principle. The differences in test points and satisfaction between groups are analyzed using Student's T-test, and the differences in proportions are analyzed using Chi-square test. Statistical significance is set at p<0.05. Analysis are performed using Rv3.6.1 and SPSS.25 statistical softwares.

ELIGIBILITY:
Inclusion Criteria:

* Patients who met ESPGHAN criteria for AGE: decreased stool consistency and/or increased evacuation frequency during a period <7 days, associated or not to fever or vomiting.
* Patients accompanied by a usual caregiver.

Exclusion Criteria:

* Patients with severe dehydration
* Patients with chronic comorbidities needing special instructions (i.e. neurologic, respiratory or cardiologic)
* Patients whose caregivers were not able to communicate in Spanish
* Patients who were admitted for hospitalization.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 139 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in test score | From 3 days to 10 days after first emergency care visit
  We calculated the difference between the score obtained in the initial test and the score obteined in the follow-up test and compared between groups. Scores are based on a 5-question test, minimum score is 0 points and maximum score (best score) is 5 points

SECONDARY OUTCOMES:
Number of caregivers getting a total score of 5 points | From 3 days to 10 days after first emergency care visit
  We measured how many caregivers got a 5-score (perfect) in the follow up test after interventions, and compared between groups
Rate of return visits | 72 hours from from the first emergency care visit
  We asked caregivers whether they had returned to emergency care or to pediatric outpatient clinics for the same problem after the first visit.
Satisfaction score with the information received | From 3 days to 10 days after first emergency care visit
  We asked caregivers to give a score between 1 and 10 (1 very unsatisfied, 10 very satisfied) regarding how useful they felt that the information given to them had been.

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Solís, M.D., Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (1):
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD are available under request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available as soon as published. It will be available for 20 years (year 2040)
Access Criteria: Investigators with research accepted by a research ethics committee conducting research in this area.

DOCUMENTS (2):
  • Informed Consent Form (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT04463355/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT04463355/Prot_SAP_001.pdf